CLINICAL TRIAL: NCT04473066
Title: Long-term Follow-up of Children With Obstructive Sleep Apnoea Treated With Adenotonsillectomy: Cardiovascular Perspectives
Brief Title: Long-term Follow-up of Children With OSA Treated With AT
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun-Ting AU, PhD, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HMRF-07181276
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea, adenotonsillectomy, cardiovascular
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adenotonsillectomy (AT): Children diagnosed with moderate-to-severe OSA (OAHI ≥3/h) and tonsillar hypertrophy (tonsil grade ≥2) at the age of 5-12 years old and underwent AT since 2012.
  Interventions: Procedure: Adenotonsillectomoy +/- turbinate reduction
- Refused AT: Children diagnosed with moderate-to-severe OSA and tonsillar hypertrophy but refused AT in the same period.
- Normal control: Children reported to have no habitual snoring (less than 3 nights per week) and confirmed to have no OSA (OAHI <1/h) by overnight sleep study in the same period.

INTERVENTIONS:
Procedure: Adenotonsillectomoy +/- turbinate reduction — Tonsillectomies were performed by bipolar electrocautery while adenoidectomies were done by monopolar suction diathermy. Turbinate reduction (by either submucosal bipolar diathermy or radiofrequency) would be offered if the subject had on-going history of allergic rhinitis and examination revealed at least grade II turbinate hypertrophy. (Grade I = no turbinate hypertrophy; Grade II = turbinate hypertrophy without touching the septum; Grade III = turbinate hypertrophy touching the septum).
  Groups: Adenotonsillectomy (AT)

SUMMARY:
Objectives: To assess the cardiovascular outcomes of children with obstructive sleep apnoea (OSA) at a mean of 5 years after they had undergone adenotonsillectomy (AT), compared to OSA children who did not undergo AT, and normal controls without OSA.

Hypothesis to be tested: (1) children with OSA underwent AT would have lower cardiovascular risks, namely lower ambulatory blood pressure (ABP), better cardiac function, lower carotid intima-media thickness (CIMT) and lower carotid arterial thickness when compared to those with OSA but did not undergo AT, and that (2) children with OSA, despite treatment with AT, would have higher cardiovascular risks than non-OSA controls. Design: A two-centre prospective case-control follow-up study Subjects: Potential subjects for this follow-up study have been identified from two local hospitals, Prince of Wales and Kwong Wah Hospitals. AT-treated group (n=90) - Children had moderate-to-severe OSA (obstructive apnoea hypopnoea index (OAHI) >=3 events/h) and underwent AT when they were aged 5-12 years. Refused AT group (n=45) - Children had moderate-to-severe OSA but refused AT. Non-OSA control group (n=45) - Non-snoring controls with OAHI <1 event/h . Main outcome measures: 24-hour ABP, cardiac function measured by echocardiography, CIMT and carotid arterial stiffness.

Data analysis: Apart from group comparisons, multiple linear regression and logistic regression analysis will also be used to examine whether cardiovascular outcomes are associated with AT, pre- and post-AT OAHI while adjusted for confounders.

Expected results: AT improves cardiovascular outcomes of children with OSA. However they still had higher cardiovascular risks than normal controls even after AT.

DETAILED DESCRIPTION:
Aims and Hypotheses to be Tested:

The primary aim of this study is to assess cardiovascular outcomes of children with OSA at a mean of 5 years after they had undergone AT, compared to OSA children without surgical treatment and children without OSA. The secondary aim is to explore factors associated with cardiovascular outcomes in subjects with OSA after AT.

We hypothesise that (1) children with OSA underwent AT would have lower cardiovascular risks, namely lower ABP, better cardiac function, lower carotid intima-media thickness (CIMT) and lower carotid arterial stiffness when compared to those with OSA but did not undergo AT, and that (2) children with OSA, despite treatment with AT, would have higher cardiovascular risks than non-OSA controls.

Study design: A two-centre prospective case-control follow-up study.

Sample size estimation:

We have conducted a pilot study to compare 12 children with residual OSA after AT (defined as post-AT OAHI >=3/h) and 12 age-, sex- and BMI-matched non-snoring controls. The results showed that children with residual OSA had a higher nighttime systolic BP (NSBP) than non-snoring controls (98.9 c.f. 95.6 mm Hg, mean difference = 3.35 mmHg, common SD = 6.54 mmHg, effect size = 0.51). We have a total of 130 subjects with moderate-to-severe OSA who had undergone AT. As the main aim of this study is to assess the treatment effects of AT, we will try to recruit as many AT-treated subjects as possible. Assuming a response rate of 70%, 90 subjects will be recruited. If 45 normal controls were also recruited (case/control ratio = 2:1), the study would provide a power of 87% to detect the difference with a 5% type I error rate. The minimum number of subjects required to detect the difference with an 80% power and a 5% type I error rate are 72 cases and 36 controls if the case/control ratio is 2:1. A sample size of 90 AT-treated subjects will also provide an 80% power to detect the potential effects of pre-AT OAHI and follow-up OAHI on cardiovascular outcomes with medium effect size (assuming a partial R-squared of 0.1), while adjusted for age, sex and BMI in multiple linear regression model within the AT group.

Besides, we have also conducted a separate pilot study comparing a group of 18 children with moderate-to-severe OSA treated with AT and a group of 18 age-, sex- and BMI-matched children with similar OSA severity without AT. The results showed that the nighttime systolic BP in the AT group was reduced by a mean of 2.3 mmHg at a 9-month follow-up visit, whereas the non-AT group had an increase in nighttime systolic BP by a mean of 2.3 mmHg (mean difference = 4.52 mmHg, common SD = 7.34 mmHg, effect size = 0.62). We have a total of 63 candidates for AT who had refused to undergo AT. Assuming a response rate of 70%, 45 subjects will be recruited. A total of 90 cases (AT-treated) and 45 controls (refused AT) provides a power of 95% to detect the expected difference with a type I error rate of 5%. The minimum number of subjects required to detect the difference with an 80% power and a 5% type I error rate are 50 cases and 25 controls if the case/control ratio is 2:1. All sample size and power calculations were done using G*Power (Version 3.1.9.2).

Our target is to recruit a total of 180 subjects, comprising of 90 OSA subjects treated with AT, 45 non-snoring controls and 45 OSA subjects without AT for this follow-up study. We are confident to recruit the target number of subjects as we have been following up the OSA patients regularly in out-patient clinic and we also have a sufficient amount of normal control subjects for matching and recruitment.

Methods:

All participants will have to visit our unit once to undergo anthropometric measurement, overnight polysomnography (PSG), 24-hour ABPM, echocardiographic and arterial assessments. They will be arranged to come to our sleep laboratory at around 9 am in the morning. Twenty-four hour ABPM will be started after resting for 10 minutes upon arrival. Echocardiographic and arterial assessments will be subsequently arranged. They will stay until the next morning after completion of overnight sleep study and 24-h ABPM. For those who are reluctant to complete the whole study protocol, especially for control subjects who may not be willing to stay overnight for the sleep study, their symptoms will be documented by a self- or parent-report questionnaire (appendix 2), and they will have to come to our unit to undergo all the cardiovascular assessments and take the ABP monitor back home and return to us the next day when the 24-h monitoring is completed. Those failed to complete all the outcome assessments will be excluded.

Data processing and analysis:

The AT-treated group will be compared to the refused AT group and the non-snoring controls to assess the between-group differences in various cardiovascular outcomes. Student's t tests, Mann-Whitney U tests and chi-square tests will be used for the comparisons of normally distributed, non-normally distributed and categorical data, respectively. Linear and logistic regression analysis will be used to test whether OSA severity at baseline and follow-up and AT are associated with continuous (e.g. CIMT) and binary (e.g. hypertension) cardiovascular outcomes, respectively, while adjusting for age, gender and body size. Subgroup analysis will also be performed within the AT-treated group to explore factors associated with cardiovascular outcomes after AT. Particularly, the association of pre-AT and follow-up OAHI with various cardiovascular outcomes will be tested. Significance level will be set as 5%. All the analyses will be performed using the statistical software packages SPSS (SPSS Inc., Chicago, Illinois, USA).

ELIGIBILITY:
General inclusion criteria:

* Participants and their parents must understand Chinese;
* Aged 5-12 years at diagnosis.

Inclusion criteria for AT group:

* Previously diagnosed with moderate-to-severe OSA (OAHI ≥3/h);
* Tonsillar hypertrophy (tonsil grade ≥2);
* Underwent AT.

Inclusion criteria for Refused AT group:

* Previously diagnosed with moderate-to-severe OSA (OAHI ≥3/h);
* Tonsillar hypertrophy (tonsil grade ≥2);
* Refused AT.

Inclusion criteria for Normal Control group:

* Previously confirmed to have no OSA (OAHI <1/h);
* Reported to have no habitual snoring (less than 3 nights per week).

Exclusion Criteria:

* Additional upper airway surgery other than the one done at baseline visit;
* Known medical conditions that affects the cardiovascular system;
* Any use of medications that alters cardiovascular system.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Potential subjects for this follow-up study have been identified from two local hospitals, Prince of Wales Hospital and Kwong Wah Hospital. Since 2012, a total of 193 candidates for AT have been identified, of whom 130 underwent AT, whilst the remaining 63 (33%) preferred more conservative treatment. Non-snoring controls have been identified in several of our previous studies that involved normal controls, including OSA family study and primary snoring follow-up study, and an ongoing study which validates a prediction model for childhood OSA. At the time of writing, a total of 258 non-snoring controls have been identified from various studies since 2012.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
24-hour ambulatory blood pressure measurements | At a mean of 5 years after intervention
  All subjects will undergo 24-hour ABPM on the same day as PSG. An validated oscillometric monitor (SpaceLabs 90217, SpaceLabs Medical, Redmond, Washington, USA) will be used. Systolic, diastolic and mean arterial BP will be measured every half-hourly during the period starting from 2200h to 0800h (nighttime period) and every 15 minutes outside of this period (daytime period). The exact cutoff time dividing wake and sleep BP will be defined individually according to the concurrent sleep study. The proper cuff (cuff size should have a bladder width that is approximately 40% of the arm circumference midway between the olecranon and the acromion precesses) is chosen according to the length of the arm of the subject and it will be placed in the nondominant arm of the child.
Cardiac function | At a mean of 5 years after intervention
  Based on M-mode assessment of the parasternal short-axis view at the mid-ventricular level, the left ventricular (LV) wall thickness and interventricular septum thickness at end-diastole will be determined. The fractional shortening and LV mass will be calculated according to standard formulae. The pulmonary arterial pressure will be estimated using the tricuspid regurgitation (TR) jet and pulmonary artery acceleration time.
  Tissue Doppler echocardiography will be performed with the sample volume positioned at the basal right ventricular (RV) and LV free-wall and interventricular septal annular junction.
  Speckle-tracking echocardiography will be performed for evaluation of myocardial deformation.
Carotid intima-media thickness | At a mean of 5 years after intervention
  The intima-media thickness (IMT) of the right and left common carotid arteries far wall at about 10 mm proximal to the carotid bulb will be measured using a 7 to 15-MHz high frequency linear-array transducer. Intima-media thickness of bilateral common carotid arteries will be automatically measured with electronic callipers. The average of three measurements from each side will be used for further analyses.
Arterial stiffness | At a mean of 5 years after intervention
  Carotid arterial stiffness of the right and left carotid arteries at about 10 mm proximal to the carotid bulb will be determined by calculation of the stiffness index.[41] Measurements of the end-diastolic (Dd) and systolic (Ds) diameters will be obtained between the far wall and near wall intima. For each systolic and diastolic diameter, three measurements from each side will be averaged and the means will be subsequently used in the calculation of the stiffness index as ln (SBP/DBP)/(ΔD/D), where SBP is right brachial systolic blood pressure, DBP is right brachial diastolic blood pressure, ΔD is the difference between systolic and diastolic diameters, and D is the diastolic diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Ting Au, PhD, Principal Investigator — junau@cuhk.edu.hk
Locations (2):
- Hong Kong (2):
  - Department of Paediatrics, Kwong Wah Hospital, Hong Kong, Kowloon
  - Department of Paediatrics, The Chinese University of Hong Kong, Shatin

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified individual participant data that underlie the results in this article (text, tables and figures) will be made available, in addition to study protocol. The data will be made available upon publication to researchers who provide a methodologically sound proposal for individual participant data meta-analysis.